CLINICAL TRIAL: NCT02213224
Title: Evaluation of Perindopril and Telmisartan for the Treatment of Nonalcoholic Fatty Liver Disease: A Randomized Controlled Trial
Brief Title: Perindopril and Telmisartan for the Treatment of Nonalcoholic Fatty Liver Disease
Acronym: NF-NAFLD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAFLD20140805
Record Dates: First submitted 2014-08-06; First posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD)
Keywords: Perindopril,Telmisartan, Efficacy, NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Perindopril; Telmisartan; Amlodipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Perindopril (Experimental): Perindopril 4mg qd taken in the morning;
  Interventions: Drug: Perindopril
- Telmisartan (Experimental): Telmisartan 80mg qd taken in the morning;
  Interventions: Drug: Telmisartan
- Amlodipine (Placebo Comparator): Amlodipine；5mg qd taken in the morning.
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Perindopril — Perindopril is a kind of angiotensin converting enzyme inhibitors (ACEIs) which has been considered as the first-line drugs for the treatment of hypertension and has been proved safe during the widespread use.
  Other Names: Perindopril; brand name: Acertil, serial number:H20034053
  Arms: Perindopril
Drug: Telmisartan — Telmisartan is a kind of angiotensin receptor blockers (ARBs) which has also been considered as the first-line drugs for the treatment of hypertension and has been proved safe during the widespread use.
  Other Names: Telmisartan; brand name: Micardis, serial number:J20090089
  Arms: Telmisartan
Drug: Amlodipine — Amlodipine is also a kind of widely used first-line drugs for the treatment of hypertension, and there is no evidence showing that it is effective for NAFLD.
  Other Names: Amlodipine；5mg qd taken in the morning.
  Arms: Amlodipine

SUMMARY:
The aim of this current study was to assess the therapeutic effects of perindopril and telmisartan for hypertensive patients with NAFLD and make comparison between the therapeutic effects of these two kind of drugs.

This study is a randomized parallel control clinical trial which would be carried out in Nanfang Hospital, Southern Medical University.

About one hundred and eighty patients would be randomly assigned to perindopril,telmisartan and amlodipine three groups.

DETAILED DESCRIPTION:
Inclusion criteria:

18-70 years old patients who were diagnosed with mild-moderate hypertension and NAFLD; The patients did not take ACEIs or ARBs drugs six weeks before the inclusion; Patients agreed to participate in the trial and signed the informed consent.

Exclusion criteria:

There are no coexisting causes for chronic liver disease, such as viral, alcoholic,drug-induced and autoimmune liver diseases; Patients with diabetes mellitus; Patients with serious primary diseases; Patients with mental disorder or can not take the medicine regularly; Pregnancy and nursing mothers; Allergic constitution or intolerance to ACEIs or ARBs drugs. Outcome measures include Cap value of FibroScan,angiotensin II,IL-18，IL-1β,aminotransferase,lipids and HOMA-IR.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old patients who were diagnosed with mild-moderate hypertension and NAFLD;
* The patients did not take ACEIs or ARBs drugs six weeks before the inclusion; Patients agreed to participate in the trial and signed the informed consent.

Exclusion Criteria:

* There are no coexisting causes for chronic liver disease, such as viral, alcoholic,drug-induced and autoimmune liver diseases;
* Patients with diabetes mellitus; Patients with serious primary diseases; Patients with mental disorder or can not take the medicine regularly;
* Pregnancy and nursing mothers;
* Allergic constitution or intolerance to ACEIs or ARBs drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Cap value of FibroScan （dB/m） | 48 weeks after the treatment
  FibroScan examination would be performed in all patients 48 weeks after administration of the drugs, and Cap value of FirbroScan will be recorded.

SECONDARY OUTCOMES:
Angiotensin II | 12, 24, 48 weeks after the treatment
IL-18，IL-1β | 12, 24, 48 weeks after the treatment
aminotransferase | 12, 24, 48 weeks after the treatment
lipids | 12, 24, 48 weeks after the treatment
HOMA-IR | 12, 24, 48 weeks after the treatment
  homeostasis model assessment of insulin resistance (HOMA-IR)
computed tomography value of liver | 48 weeks after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Side Liu, MD,PhD, Principal Investigator — Department of Gastroenterology, Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China